CLINICAL TRIAL: NCT04284527
Title: Validity and Reliability of the Assessment of Physiotherapy Practice Validation as a Measure in Physiotherapy Student
Brief Title: The Assessment of Physiotherapy Practice Validation as a Measure in Physiotherapy Student
Acronym: APP
Status: Completed | Type: Observational
Sponsor: Universidad Católica San Antonio de Murcia (Other)
Responsible Party: Principal Investigator, Jasemin Todri, Principal investigator, Universidad Católica San Antonio de Murcia
Other Study IDs: 53383
Record Dates: First submitted 2020-02-24; First posted 2020-02-25 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-09

CONDITIONS: Assessment, Self; Clinical Performance
Keywords: physiotherapy; student; assesment tool
MeSH Terms: interventions — Observation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Observational study — a reliability - validity study

SUMMARY:
The objective of this study is to determine the reliability and validity of the assesment of physiotherapy practice (APP) in physiotherapy students. Concretely the study aims to verify if the APP created by the professors of specific methods of intervention in physiotherapy course is a reliable tool to evaluate student performance of history taking and physical examination in the same course.

DETAILED DESCRIPTION:
Before evaluating this scale, the investigators want to verify the effectiveness of this online practice in the COVID period by processing the Mind Genomics questionnaire.

After the fist online results of this practice evaluation the investigators have to interpret and evaluate the APP.

ELIGIBILITY:
Inclusion Criteria:

* students of specific methods of intervention in physiotherapy course
* students of Catholic University of Murcia, Spain
* with a minimum of 19 years old
* in the second course of physiotherapy

Exclusion Criteria:

* other courses participants
* professors
* segretary

Ages: 19 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Students of the specific methods of intervention in physiotherapy course of Catholic University of Murcia, Spain
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2020-03-24 (Actual); Primary Completion 2020-03-27 (Actual); Study Completion 2020-06-04 (Actual)

PRIMARY OUTCOMES:
Assessment of Physiotherapy Practice (APP) | 10 minutes
  Validity and reliability of the Assessment of Physiotherapy Practice tool with a total of 10 point valoration

CONTACTS AND LOCATIONS:
Overall Officials: Carolina Vasques Villa, PhD, Principal Investigator — UCAM Universidad Catolica de Murcia
Locations (1):
- Universidad Católica de Murcia, Murcia, Spain